CLINICAL TRIAL: NCT00322244
Title: Massage Therapy for Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Yale University (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0120020367; CORPRC #U48-CCU115802
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Massage therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Massage

INTERVENTIONS:
Procedure: Massage Therapy

SUMMARY:
The study is a randomized, controlled clinical trial that investigates the efficacy ogf massage therapy for 66 patients with pain secondary to osteoarthritis of the knee. It is a wait-list design where subjects and randomly assigned to either Group A or Group B. Group A receives two months of massage while Group B is wait-listed, receives two months of usual care. At the conclusion of the wait period, Group B receives two months of massage. In all cases, subjects continue to receive conventional medical care for their OA symptoms.

Outcome measures include a WOMAC questionnaire, a visual analog pain scale, time to walk fifty feet and range of motion of the knee (using a goniometer). A research assistant, competent in appropriate subject assessment obtains the outcome measures. Change in medication use is tracked by the use of patient diaries. Assessments of subjects, occurs at baseline, and week 8 and 16 in both the intervention and control groups.

DETAILED DESCRIPTION:
The Yale-Griffin Prevention Research Center has received funding from the Centers for Disease Control and Prevention to conduct the Complementary and Alternative Medicine (CAM) Outcomes Research Project (CORP). CORP includes a systematic review of the CAM literature and the development of pilot studies assessing selected CAM interventions. The first year efforts of the CORP research team have culminated in the selection of pilot studies involving three public health priority conditions (attention deficit hyperactivity disorder, asthma, and osteoarthritis) and common CAM interventions. A pilot study investigating the effects of a massage therapy intervention for osteoarthritis is detailed in this application.

Osteoarthritis (OA), the most common form of arthritis, is a slowly progressive degenerative disease of joint cartilage that afflicts 30 million Americans (Praemer A, Furner S, Rice D. Musculoskeletal Conditions in the United States, p 40: American Academy of Orthopaedic Surgeons, 1992). It becomes more prevalent with advancing age (Peyron JG. Osteoarthritis: The Epidemiologic ViewPoint. Clin Orthop, 213:13-19, 1986). Nearly half of America's elderly suffer from osteoarthritis, and arthritis is the most frequently reported chronic condition in the elderly (Praemer A, Furner S, Rice D. Musculoskeletal Conditions in the United States, p 36: American Academy of Orthopaedic Surgeons, 1992).

Osteoarthritis affects approximately 3 out of every 100 Americans below age 45 and more than a quarter of Americans between the ages of 45 and 64 suffer from this disabling disease (National Center for Health Statistics. Current Estimates from the National Health Interview Survey, 1988; Vital and Health Statistics. Series 10: No. 173, DHHS Pub. No. (PHS) 89-1501. Public Health Service, Hyattsville, MD, Oct. 1989; Kelsey JL, Hochberg MC. Epidemiology of Chronic Musculoskeletal Disorders. Am Rev Public Health, 91:379-401, 1988).

Osteoarthritis of the hip or knee is particularly disabling because it limits ambulation, but the affliction also strikes the hands, the spine, and the feet with the same destructive joint process (Felson DT. Epidemiology of Osteoarthritis: Prevalence and Risk Factors. Osteoarthritis Disorders, American Academy of Orthopaedic Surgeons, 1995). The endpoint of the OA disease process is total loss of joint cartilage in the affected area and the need for joint replacement.

The high prevalence of arthritis in the population is reflected in the economic burden engendered to treat those afflicted. The total cost of conventional treatments for arthritis in 1988, for example, was estimated at 54.6 billion dollars (Lazenby HC, Letsch SW. National Health Expenditures 1989; Health Care Financing Review, 12(2):1-26, 1990). Conventional treatments for OA include pain medication (NSAIDS and cox-2 inhibitors), exercises, hot/cold therapy, steroid injections and, eventually, surgery to repair the joint (Felson DT. Epidemiology of Osteoarthritis: Prevalence and Risk Factors. Osteoarthritis Disorders, American Academy of Orthopaedic Surgeons, 1995). Despite conventional treatment, OA is a progressive disease that frequently leads to chronic pain and disability.

Massage therapy is proposed as an effective treatment for diminishing the symptoms and improving the disease course of osteoarthritis. Massage therapy can accomplish these goals by increasing local circulation to the affected joint, improving the tone of supportive musculature, enhancing joint flexibility and relieving pain (J Spinal Cord Med 2001 Spring; 24(1): 54-62.).

Massage therapy has been evaluated and found to have effectiveness as an adjunct treatment for pain secondary to cancer (Effects of massage on pain intensity: analgesics and quality of life in patients with cancer pain: A pilot study of a randomized clinical trial conducted within hospice care delivery. Wilkie, DJ et al.) as well as low back pain syndrome (Preyde, M. Effectiveness of massage therapy for subacute low-back pain. Journal Burn Care & Rehab 2000; 21(3): 189-193.). It also has been shown to be beneficial for patients with chronic pain following spinal cord injury (Nayak S, Matheis RJ, Agostinelli S, Shiflett SC. The use of complementary and alternative therapies for chronic pain following spinal cord injury: a pilot survey. CMAJ 2000; 162(13): 1815-1820). In a randomized, open clinical trial, a series of classical Swedish massage therapy sessions was found to be as effective as conventional analgesic therapy for chronic rheumatic pain. (Ernst E. Complementary and alternative medicine for pain management in rheumatic disease. Current Opinion in Rheum 2002; 14:58-62). However, to date, no study has specifically evaluated the effectiveness of massage therapy for osteoarthritis.

The proposed study is a randomized, controlled clinical trial to investigate the efficacy of massage therapy for patients with pain secondary to osteoarthritis of the knee. It is a wait-list design where subjects will be randomly assigned to either Group A or Group B. Group A will receive two months of massage while Group B is wait-listed, receiving two months of usual care. At the conclusion of the wait period, Group B will receive two months of massage. In all cases, subjects will continue to receive conventional medical care for their OA symptoms.

Outcome measures will include a WOMAC questionnaire (see Appendix A), a visual analog pain scale (see Appendix B), time to walk fifty feet, and range of motion of the knee (using a goniometer). An athletic trainer, competent in appropriate subject assessment, will obtain the outcome measures (see Appendix C for data collection form). Change in medication use will be tracked by the use of patient diaries (see Appendix D). Assessment of subjects will occur at baseline, and weeks 8 and 16 in both the intervention and control groups.

The intervention will consist of one-hour massage therapy sessions as follows:

Weeks one through four: twice weekly Weeks five through eight: weekly

Initial treatments are given with greater frequency to "build a loading dose" of massage treatments, effecting a greater impact at the onset of treatment. The preponderance of published studies built in twice-weekly massage for four to five weeks at the onset of treatment (Field, T. et al. Bulimic adolescents benefit from massage therapy. Adolescence 1997 33, 131; Leivadi, S. et al. Massage therapy and relaxation effects on university dance students. Journal of Dance Medicine & Science 1999, 3, 108-112).

Nationally certified and licensed massage therapists who have graduated from an accredited school of massage therapy will give the massage therapy intervention. The therapists will follow standard Swedish full-body therapeutic massage technique. In order to minimize practitioner variability of treatment, a standardized protocol incorporating a sequence of strokes (effleurage, petrissage, tapotement) has been developed (see Appendix E). Subjects will remain supine or prone for the full hour of treatment, turning over roughly at the halfway point.

The second group will begin receiving the identical intervention after the first group has completed its treatment. Weekly phone calls to encourage the second group will be made to minimize attrition. The first group will be followed via phone interviews, with follow-up data collected until the conclusion of the study.

Subjects will be men and women with an established diagnosis of OA meeting ACR criteria, 35 years of age or greater, with a score of 4-9 on a visual analogue scale. Subjects will not be excluded based on gender or race.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically confirmed diagnosis of osteoarthritis
* 35 years of age or greater
* pre-randomization VAS score between 4 and 9

Exclusion Criteria:

* Rheumatoid, arthritis, fibromyalgia, recurrent or active pseudo-gout, cancer or other serious medical condition
* History of kidney or liver failure
* Asthma requiring steroids
* oral steroids within the last four weeks
* Intra-articular knee depo-corticosteroids within the previous 3 months
* Intra-articular hyaluronate within the previous 6 months
* Arthroscopy of the knee within the previous year
* Significant injury to the knee within the previous 6 months
* rash or open wound over the knee

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2003-01; Study Completion 2003-10

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain and functional scores
Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Range of motion
Time to walk 50 feet

CONTACTS AND LOCATIONS:
Overall Officials: Adam I. Perlman, MD, MPH, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- Saint Barnabas Ambulatory Care Center, Livingston, New Jersey, United States

REFERENCES:
- [Derived] Perlman AI, Sabina A, Williams AL, Njike VY, Katz DL. Massage therapy for osteoarthritis of the knee: a randomized controlled trial. Arch Intern Med. 2006 Dec 11-25;166(22):2533-8. doi: 10.1001/archinte.166.22.2533. PMID 17159021